CLINICAL TRIAL: NCT01854827
Title: A Phase 1/2A Trial of Intravenous Immunoglobulin (IVIG) Therapy Following Portoenterostomy in Infants With Biliary Atresia
Brief Title: Safety Study of Intravenous Immunoglobulin (IVIG) Post-Portoenterostomy in Infants With Biliary Atresia
Acronym: PRIME
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P007 PRIME; U01DK062456 (NIH)
Record Dates: First submitted 2012-09-27; First posted 2013-05-16 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Biliary Atresia
Keywords: Biliary atresia; Hepatic portoenterostomy; Intravenous immunoglobulin
MeSH Terms: conditions — Biliary Atresia | interventions — Immunoglobulins, Intravenous; Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IVIG active treatment (Experimental): Intravenous immunoglobulin (IVIG) 10% 1 gm/kg body weight/dose Day 3-5,30, 60 post HPE
  Interventions: Drug: Intravenous immunoglobulin (IVIG)

INTERVENTIONS:
Drug: Intravenous immunoglobulin (IVIG) — All participants will receive the same dose of IVIG at the same intervals in an open-label fashion as long as the subject does not have any increased risk for toxicity for any IVIG infusion. IVIG will be initiated on day 3 (up to day 5) after HPE surgery (HPE is day 0) at a dose of 1 gm/kg body weight by slow intravenous infusion over at least 4 hours. The same dose (1 gm/kg) and duration of infusion will be repeated on day 30 and day 60 after HPE.
  Other Names: Gamunex-C®; Gamunex®

SUMMARY:
The Children Liver Disease Research and Education Network (ChiLDREN) is conducting a clinical trial to determine the feasibility, acceptability, tolerability and safety profile of IVIG treatment administered to infants after hepatic portoenterostomy (HPE) for biliary atresia, as well as investigate preliminary evidence of activity and explore mechanisms of action.

DETAILED DESCRIPTION:
In this multicenter prospective phase 1/2A open label trial, the feasibility, tolerability and safety of intravenous immunoglobulin (IVIG) therapy following hepatic portoenterostomy (HPE) will be assessed in 29 infants with biliary atresia (BA), efficacy will be estimated and exploratory mechanistic research studies will be performed. After written consent is obtained from the parent or guardian, the subject will be enrolled and will receive three intravenous doses of IVIG at designated intervals over the first 60 days following HPE and will be followed for 360 days after enrollment. Blood will also be obtained during this study to assess potential mechanisms by which the IVIG may alter or reduce bile duct inflammation and injury and improve bile flow. All infants in this trial will also be treated with standardized doses of other routine standard-of-care treatments for BA during this trial (ursodeoxycholic acid, trimethoprim-sulfamethoxasole, and fat-soluble vitamin supplements). This routine clinical care will not be modified by participation in this study. Subjects in this study will not receive corticosteroid therapy for treatment of biliary atresia, as this is of unproven benefit at the present time.

ELIGIBILITY:
Inclusion Criteria:

* Infant under 120 days old with established diagnosis of BA. Subjects in this trial must start treatment within 3-5 days of the Kasai procedure and be part of a prospective study of the natural history of biliary atresia also being conducted by ChiLDREN (http://www.clinicaltrials.gov/ct/show/NCT00061828?order=3).
* Standard HPE operation has been performed for BA within the previous 3 days
* Post-conception age ≥ 36 weeks at time of enrollment
* Weight at enrolment ≥ 2000 gm
* Written informed consent to participate in the study obtained within 3 days of completion of HPE.

Exclusion Criteria:

* Laparoscopic HPE or "gall bladder Kasai" (cholecysto-portostomy) surgery was performed
* Biliary atresia splenic malformation syndrome (presence of asplenia, polysplenia or double spleen)
* History of a hypercoagulable disorder
* Renal Disease defined as serum creatinine > 1.0 mg/dl prior to enrollment or presence of complex renal anomalies found on imaging
* Evidence of congestive heart failure or fluid overload
* Presence of significant systemic hypertension for age (defined as persistent systolic blood pressure ≥112 mmHg measured on at least 3 occasions following HPE)
* Infants whose mother is known to have human immunodeficiency virus infection
* Infants whose mother is known to be serum HBsAg or hepatitis C virus antibody positive
* Previous treatment with intravenous immunoglobulin therapy or corticosteroid therapy
* Previous treatment with any other investigational agent
* History of allergic reaction to any human blood product infusion
* Infants with other severe concurrent illnesses, such as neurological, cardiovascular, pulmonary, metabolic, endocrine, and renal disorders, that would interfere with the conduct and results of the study
* Any other clinical condition that is a contraindication to the use of IVIG

Ages: 3 Days to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Sokol, MD, Study Chair — Children's Hospital Colorado; Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Disease (NIDDK); Averell Sherker, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Disease (NIDDK)
Locations (7):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital at Pittsburgh, Pittsburgh, Pennsylvania
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Mack CL, Spino C, Alonso EM, Bezerra JA, Moore J, Goodhue C, Ng VL, Karpen SJ, Venkat V, Loomes KM, Wang K, Sherker AH, Magee JC, Sokol RJ; The ChiLDReN Network. A Phase I/IIa Trial of Intravenous Immunoglobulin Following Portoenterostomy in Biliary Atresia. J Pediatr Gastroenterol Nutr. 2019 Apr;68(4):495-501. doi: 10.1097/MPG.0000000000002256. PMID 30664564
- See also: Click here for more information about the Children Liver Disease Research and Education Network (ChiLDREN) — https://childrennetwork.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IVIG Active Treatment
Started | 30
Completed | 29
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: MITT (Modified Intent-to-Treat) defined as all patients receiving at least one does of IVIG and maintaining eligibility throughout the trial.
Groups:
- IVIG Active Treatment: Intravenous Immunoglobulin (IVIG) active treatment for infants with biliary atresia
Arm/Group | IVIG Active Treatment
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: Days] | 60.0 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 9
  Ethnicity: Non-Hispanic | 20
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 7
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of IVIG Treatment
Description: Percentage of subjects for whom administration of IVIG is feasible, defined as the successful administration (at least 80% of each dose) of all 3 doses of IVIG
Time Frame: 60 days post-HPE
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG Active Treatment
Number analyzed (Participants) | 29
Participants | 23
Statistical Analysis 1: Comparison: IVIG Active Treatment; Test type: Superiority — Percent was evaluated relative to 80% where statistical superiority was demonstrated if the one-sided, 90% Clopper-Pearson lower confidence bound was > 80%; Percent of patients = 79.3, 90% CI 1-sided [lower limit 63.2]; The lower bound of the 90% Clopper-Pearson confidence interval was < 80%, therefore the study failed to achieve the feasibility definition stated in the protocol

2. Primary Outcome: Acceptability of IVIG
Description: Percentage of subjects for whom the study is acceptable, defined as the ability of the subject's family or guardian to allow intravenous line placements, blood draws, and other study procedures for the study subjects.
Time Frame: 60 days post-HPE
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG Active Treatment
Number analyzed (Participants) | 29
Participants | 23
Statistical Analysis 1: Comparison: IVIG Active Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Percent of patients = 79.3, 90% CI 1-sided [lower limit 63.2]; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Serious Adverse Events
Description: Percentage of subjects with any serious adverse events (SAEs) prior to liver transplant
Time Frame: 360 days post-HPE
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG Active Treatment
Number analyzed (Participants) | 29
Participants | 26
Statistical Analysis 1: Comparison: IVIG Active Treatment; Test type: Other — Percents with serious AEs prior to liver transplant were calculated, along with one-sided 90% Clopper-Pearson confidence interval lower bounds; Percent of patients = 89.7, 90% CI 1-sided [lower limit 75.4]

4. Primary Outcome: Level 3-5 Toxicity
Description: Percentage of subjects with any level 3, 4, or 5 toxicity (per NCI CTEP grading system)
Time Frame: 360 days post-HPE
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG Active Treatment
Number analyzed (Participants) | 29
Participants | 26
Statistical Analysis 1: Comparison: IVIG Active Treatment; Test type: Other — Percent of patients with level 3-5 toxicity are presented along with one-sided 90% Clopper-Pearson confidence interval lower bound; Percent of patients = 89.7, 90% CI 1-sided [lower limit 75.4]

5. Primary Outcome: Adverse Events
Description: Percentage of subjects with other expected adverse events
Time Frame: 360 days post-HPE
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG Active Treatment
Number analyzed (Participants) | 29
Participants | 8
Statistical Analysis 1: Comparison: IVIG Active Treatment; Test type: Other — Percent of patients with other expected AEs are presented along with one-sided 90% Clopper-Pearson confidence limit lower bound; Percent of patients = 27.6, 90% CI 1-sided [lower limit 14.5]

6. Secondary Outcome: Good Bile Drainage at 90 Days Post-HPE
Description: Percentage of subjects who survive 90 days after HPE with both their native liver and serum total bilirubin <1.5 mg/dL at 90 days after HPE
Time Frame: 90 days post-HPE
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG Active Treatment
Number analyzed (Participants) | 29
Participants | 11
Statistical Analysis 1: Comparison: IVIG Active Treatment; IVIG was compared to the historical placebo control from the START study (n=64): PMID: 24794368 NCT00294684; Test type: Superiority — One-sided testing for superiority of IVIG to historical control; p = 0.5486, Regression, Logistic; Odds Ratio (OR) = 0.67, 90% CI 1-sided [upper limit 2.38]

7. Secondary Outcome: Good Bile Drainage at 180 Days Post-HPE
Description: Percentage of subjects who survive 180 days after HPE with both their native liver and serum total bilirubin <1.5 mg/dL at 180 days after HPE
Time Frame: 180 days post-HPE
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG Active Treatment
Number analyzed (Participants) | 29
Participants | 14
Statistical Analysis 1: Comparison: IVIG Active Treatment; IVIG was compared for superiority to the historical control of START study placebo (N=64). PMID: 24794368 NCT00294684; Test type: Superiority — One-sided testing for superiority of IVIG relative to historical control; p = 0.8455, Regression, Logistic; Odds Ratio (OR) = 0.33, 90% CI 1-sided [upper limit 1.22]

8. Secondary Outcome: Good Bile Drainage at 360 Days Post-HPE
Description: Percentage of subjects who survive 360 days after HPE with both their native liver and serum total bilirubin <1.5 mg/dL at 360 days after HPE
Time Frame: 360 days post-HPE
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG Active Treatment
Number analyzed (Participants) | 29
Participants | 7
Statistical Analysis 1: Comparison: IVIG Active Treatment; IVIG was compared for superiority to the historical START placebo control (N=64); Test type: Superiority — One-sided; p = 0.8431, Regression, Logistic — One-sided; Odds Ratio (OR) = 0.29, 90% CI 1-sided [upper limit 1.24]

9. Secondary Outcome: Transplant-free Survival
Description: Percentage of subjects who survive with their native liver at 360 days after HPE.
Time Frame: 360 days post-HPE
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG Active Treatment
Number analyzed (Participants) | 29
Participants | 17
Statistical Analysis 1: Comparison: IVIG Active Treatment; K-M estimates for survival for IVIG vs the historical START placebo control are provided, along with one-sided 90% upper bounds of the confidence intervals; Test type: Superiority — One-sided for IVIG superior to historical START placebo control. PMID: 24794368 NCT00294684; Risk Difference (RD) = -11.9, 90% CI 1-sided [upper limit 2.1]

10. Secondary Outcome: Circulating Regulatory T-Cells, Inflammatory Cytokines, and Specific Autoantibodies.
Description: Percentage and absolute number of Tregs (CD4+CD25+FoxP3+), CD3/4 T cells, CD3/8 T cells, NK cells (CD56), NK T cells (CD3/56), CD19/20 B cells, macrophages (CD14/11b), and neutrophils; plasma levels of anti-enolase antibody; and plasma cytokine levels (Th1/Th2 multiplex and IL17)
Time Frame: Over 360 days after HPE
Reporting Status: Not Posted, anticipated posting 2019-10

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment into the study until the earlier of the Day 365 visit or withdrawal from the study.
Arm/Group | IVIG Active Treatment
All-Cause Mortality (participants affected / at risk) | 1/29
Serious Adverse Events (participants affected / at risk) | 26/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG Active Treatment (N=29)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 3 (3)
Hepatic (Hepatobiliary disorders) | 12 (20)
Immunological (Immune system disorders) | 3 (3)
Infectious (Infections and infestations) | 21 (63)
Metabolic (Metabolism and nutrition disorders) | 1 (1)
Neoplastic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Nutritional (Metabolism and nutrition disorders) | 10 (13)
Surgical (Surgical and medical procedures) | 2 (2)
Post Operative Liver Transplant (Surgical and medical procedures) | 12 (12)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG Active Treatment (N=29)
Constipation (Renal and urinary disorders) | 4 (6)
Acholic Stools (Renal and urinary disorders) | 14 (22)
Allergic Reaction (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 5 (8)
Ascites (Hepatobiliary disorders) | 16 (21)
Cold Systems (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Other (General disorders) | 28 (168)
Decreased Feeding (Metabolism and nutrition disorders) | 12 (13)
Dehydration (General disorders) | 1 (1)
Diaper Rash (Skin and subcutaneous tissue disorders) | 9 (11)
Diarrhea (Renal and urinary disorders) | 12 (17)
Difficulty Breathing (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4)
Edema (Skin and subcutaneous tissue disorders) | 1 (1)
Elevated Bilirubin (Hepatobiliary disorders) | 7 (10)
Elevated INR (Hepatobiliary disorders) | 6 (7)
Elevation in AST and/or ALT (Hepatobiliary disorders) | 2 (2)
Elevation in Systolic BP > 112 (Cardiac disorders) | 7 (9)
Emesis (Gastrointestinal disorders) | 11 (21)
Feeding Intolerance (Metabolism and nutrition disorders) | 1 (1)
Fever (Infections and infestations) | 18 (51)
Fussiness (Psychiatric disorders) | 3 (7)
Gastrointestinal (Gastrointestinal disorders) | 3 (3)
Hepatic (Hepatobiliary disorders) | 13 (24)
Hypotension (Cardiac disorders) | 1 (1)
Immunological (Immune system disorders) | 3 (3)
Inadequate wait gain (Metabolism and nutrition disorders) | 2 (2)
Increased PT/INR (Hepatobiliary disorders) | 2 (3)
Increased Sleepiness (General disorders) | 7 (8)
Infectious (Infections and infestations) | 21 (63)
Irritability (Psychiatric disorders) | 10 (19)
Jaundice (Renal and urinary disorders) | 9 (15)
Metabolic (Metabolism and nutrition disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neoplastic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Nutritional (Metabolism and nutrition disorders) | 10 (13)
Oral Thrush (General disorders) | 3 (4)
Otitis Media (Infections and infestations) | 3 (5)
Poor Weight Gain (Metabolism and nutrition disorders) | 11 (11)
Post Operative Liver Transplant (Surgical and medical procedures) | 12 (12)
Pruitis (Skin and subcutaneous tissue disorders) | 6 (7)
RSV (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 5 (8)
Reflux (Gastrointestinal disorders) | 4 (5)
Surgical (Surgical and medical procedures) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Vomitting (Gastrointestinal disorders) | 14 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No